CLINICAL TRIAL: NCT04473729
Title: Improving Perception of Speech in Noise in Children With Communication Disorders
Acronym: L2F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smarty Ears (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Southern Connecticut State University (Unknown); Haskins Laboratories (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Listening2Faces; 3R43DC017405-01A1S1 (NIH)
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Speech Perception
Keywords: ASD; speech in noise; Hearing Loss; speech-to-noise ratio
MeSH Terms: conditions — Hearing Loss | interventions — Noise

STUDY DESIGN:
Intervention Model Description: The model is ABA design, that is participants get an initial, pre-treatment noise assessment, then get individualized training, then get a post-noise assessment. This is designed to look for change from baseline after training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Children with an autism spectrum disorder (Experimental): The intervention as described above with children with an ASD.
  Interventions: Other: Audiovisual speech training in noise for children
- Children with Hearing Loss (Experimental)
  Interventions: Other: Audiovisual speech training in noise for children
- Typically developing children with normal hearing acuity (Experimental)
  Interventions: Other: Audiovisual speech training in noise for children

INTERVENTIONS:
Other: Audiovisual speech training in noise for children — Children will participate in listening training in the form of an iPad app

SUMMARY:
Smarty Ears has developed a prototype of an innovative therapeutic training system to improve speech perception in noise by training children on interrupted noise (which has silent intervals that allow for fragments of the target to be heard). The study will attempt to validate the technology and gather initial design feedback from clinicians and caregivers and from children with ASD and HL.

DETAILED DESCRIPTION:
Recent evidence indicates that listening in interrupted noise can provide perceptual benefits, such as remapping the auditory environment and learning to use acoustic cues. The developed technology, uses adaptive listening training that automatically increases noise level difficulty as performance improves, and includes age appropriate rewards to maintain interest. The mobile app includes an initial and final screening, a training system that administers training via the child's own mobile device, and detailed performance dashboard. The study will attempt to validate the technology by gathering feedback from clinicians and caregivers and from children with ASD and HL.

ELIGIBILITY:
Inclusion Criteria:

* For all children: normal or corrected to normal vision.
* For children with typical development normal or corrected to normal vision + normal hearing.
* For children with HL Children must have at least one year experience with amplification (i.e Hearing aids) and no threshold> 70 dB.

Exclusion Criteria:

* To participate, all children must be able to comply with directions and engage in tasks that require some expressive language response on the language and cognitive measures (i.e. children who are considered to be in the "word combinations" or "sentences expressive language" phase; Tager-Flusberg et al., 2009).

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Daily training performance | 5 days a week for 4 weeks (30 minutes/day)
  Daily performance level based on words correct as a function of SNR and the average SNR over the course of training for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Fernandes, M.S, Principal Investigator — Smarty Ears
Locations (2):
- United States (2):
  - Southern Connecticut State University, New Haven, Connecticut
  - Hampton University, Hampton, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Irwin J, Preston J, Brancazio L, D'angelo M, Turcios J. Development of an audiovisual speech perception app for children with autism spectrum disorders. Clin Linguist Phon. 2015 Jan;29(1):76-83. doi: 10.3109/02699206.2014.966395. Epub 2014 Oct 14. PMID 25313714
- [Result] Irwin JR, Tornatore LA, Brancazio L, Whalen DH. Can children with autism spectrum disorders "hear" a speaking face? Child Dev. 2011 Sep-Oct;82(5):1397-403. doi: 10.1111/j.1467-8624.2011.01619.x. Epub 2011 Jul 25. PMID 21790542
- [Result] Irwin JR, Brancazio L. Seeing to hear? Patterns of gaze to speaking faces in children with autism spectrum disorders. Front Psychol. 2014 May 8;5:397. doi: 10.3389/fpsyg.2014.00397. eCollection 2014. PMID 24847297
- See also: Link to Small Business/PI on study — http://www.smartyearsapps.com